CLINICAL TRIAL: NCT07200817
Title: Comparison Between Neutrophils to Lymphocytes and Platelets Ratio, Procalcitonin, and Total Leucocytic Count as Indicators of Prognostic Outcome in Septic Patients in the Intensive Care Unit.
Brief Title: Neutrophils to Lymphocytes and Platelets Ratio, Procalcitonin, and Total Leucocytic Count as Indicators of Prognostic Outcome in Septic Patients in the Intensive Care Unit.
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, MICHAEL GAMAL SAMAAN FARAG, Assistant Lecturer of Anesthesiology, Intensive Care and Pain Management, Faculty of Medicine, Ain Shams University, Egypt., Ain Shams University
Other Study IDs: FMASU MD224/2024
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Neutrophils to Lymphocytes; Platelets; Procalcitonin; Total Leucocytic Count; Prognostic Outcome; Septic Patients; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Septic patients (under the third international consensus definitions of sepsis and septic shock)
  Interventions: Diagnostic Test: Neutrophils to Lymphocytes and Platelets ratio (N/LP)

INTERVENTIONS:
Diagnostic Test: Neutrophils to Lymphocytes and Platelets ratio (N/LP) — The Neutrophils to Lymphocytes and Platelets ratio (N/LP) will be measured

SUMMARY:
This study aims to compare Neutrophil to Lymphocyte and Platelet Ratio, Procalcitonin, and Total Leucocyte Count as indicators of prognostic outcome in septic patients in the intensive care unit.

DETAILED DESCRIPTION:
Sepsis affects more than 30 million people annually worldwide and is one of the significant causes of death in critical patients worldwide. Any infected person can potentially develop sepsis, and the incidence of sepsis is as high as 1-2% of all hospitalized patients.

Many potential sepsis biomarkers have been proposed, procalcitonin (PCT) and C-reactive protein (CRP) being the most frequently studied.

The ratio of neutrophils to lymphocytes and platelets (N/LP) is a low-cost measure that can be obtained through routine blood tests and is often used to reflect the body's inflammatory state.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 years old.
* Both sexes.
* Septic patients (under the third international consensus definitions of sepsis and septic shock).

Exclusion Criteria:

* Pregnancy
* Malignancy
* On immunosuppressive therapy
* Hematological Disorders
* Major Trauma
* Major Burns
* Child-Pugh Class C Liver Cirrhosis
* On Hemodialysis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective observational study will be conducted at Ain Shams University Hospital, Cairo, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
Levels of Neutrophils to Lymphocytes and Platelets ratio | 28 days post-procedure
  The ratio of neutrophils to Lymphocytes and Platelets in relation to 28-day mortality among septic patients will be recorded.

SECONDARY OUTCOMES:
Procalcitonin (PCT) | 28 days post-procedure
  Procalcitonin (PCT) in relation to 28day mortality among septic patients will be recorded.
Total Leukocytic Count (TLC) | 28 days post-procedure
  Total Leukocytic Count (TLC) in relation to 28day mortality among septic patients will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.